CLINICAL TRIAL: NCT00924534
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Group Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SLV337 in Patients With Type 2 Diabetes on Metformin Monotherapy
Brief Title: A Safety PK/PD Study of SLV337 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Products (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S337.2.001; 2009-011589-27 (EudraCT Number)
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; interventional; placebo; controlled; PK; PD; safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: SLV337
- 3 (Experimental)
  Interventions: Drug: SLV337
- 4 (Experimental)
  Interventions: Drug: SLV337

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 1
Drug: SLV337 — SLV337 400 mg/day
  Arms: 2
Drug: SLV337 — SLV337 800 mg/day
  Arms: 3
Drug: SLV337 — SLV337 1400 mg/day
  Arms: 4

SUMMARY:
The purpose of this study is to assess safety, tolerability, pharmacokinetics and pharmacodynamics of SLV337 in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria Type 2 diabetes ,stable dose of Metformin,HbA1c >= 7%, but < 9% Exclusion Criteria Type 1 diabetes mellitus, Body Mass Index (BMI) >40.0 kg/m2, evidence of unstable cardiovascular diseases, NYHA class I to IV, ALT > 1.5 times UNL, creatinine clearance <60 mL/min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in alanine amino transferase level to Day 35 | 35 days
Change from baseline in Creatinine level to Day 35 | 35 days
Change from baseline in the count of Red blood cells to Day 35 | 35 days
Change from baseline in White blood cells count to Day 35 | 35 days
Change from baseline in Creatinine kinase level to Day 35 | 35 days

SECONDARY OUTCOMES:
Change from baseline in Fasting plasma glucose level to Day 28 | 28 days
Change from baseline in Adiponectin level to Day 28 | 28 days
Change from baseline in Triglycerides level to Day 28 | 28 days
Change from baseline in High density lipoprotein cholesterol level to Day 28 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Francis Roy, MS, Study Director — Abbott Products
Locations (12):
- Bulgaria (4):
  - Site Reference ID/Investigator# 54183, Dimitrovgrad
  - Site Reference ID/Investigator# 54182, Pleven
  - Site Reference ID/Investigator# 44722, Plovdiv
  - Site Reference ID/Investigator# 44723, Sofia
- Poland (5):
  - Site Reference ID/Investigator# 44725, Lubin
  - Site Reference ID/Investigator# 44724, Puławy
  - Site Reference ID/Investigator# 54185, Radzymin
  - Site Reference ID/Investigator# 44727, Ruda Śląska
  - Site Reference ID/Investigator# 54184, Wroclaw
- South Africa (3):
  - Site Reference ID/Investigator# 44728, Cape Town
  - Site Reference ID/Investigator# 44730, Cape Town
  - Site Reference ID/Investigator# 44729, Johannesburg